CLINICAL TRIAL: NCT07037108
Title: Combined Effect of Reflexology and General Stretching on Insomnia Vesomotor Symptoms and Quality of Life in Post-menopausal Women
Brief Title: Combined Effect of Reflexology and GS on Insomnia Vesomotor Symptoms and QOL in Post-menopausal Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1006
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflexology + Generalized Stretching (Experimental)
  Interventions: Combination Product: Reflexology + Generalized Stretching
- Stretching Only (Active Comparator)
  Interventions: Combination Product: Stretching Only

INTERVENTIONS:
Combination Product: Reflexology + Generalized Stretching — Participants in Group 1 received a combination of foot reflexology and generalized stretching exercises. focusing on specific reflex points related to the endocrine, nervous, and reproductive systems. Each reflexology session lasted for 20 minutes, conducted three times per week for 6 weeks.
  Arms: Reflexology + Generalized Stretching
Combination Product: Stretching Only — Generalized Stretching Only Method: Generalized Stretching Exercises Details: Participants in Group 2 received only generalized stretching exercises without any reflexology treatment. The stretching protocol included exercises for major muscle groups such as the neck, shoulders, back, hips, hamstrings, and calves. Each session will last for 20-25 minutes, which included a 5-minute warm-up, 15-20 minutes of static stretching, and a 5-minute cool-down.
  Arms: Stretching Only

SUMMARY:
The purpose of this study is to assess how reflexology and general stretching affect postmenopausal women's quality of life, vasomotor symptoms, and insomnia. Hormonal changes in postmenopausal women frequently result in hot flashes, sleep difficulties, and a general reduction in quality of life. Although non-pharmacological treatments like stretching and reflexology have demonstrated promise in treating these symptoms on their own, little study has evaluated how well they work together.

DETAILED DESCRIPTION:
Purposive sampling was used to choose postmenopausal women between the ages of 45 and 60 for a randomized controlled experiment. Participants were divided into two groups at random: the group participating in the experiment received generalized stretching exercises and reflexology, whereas the control group only received stretching or routine care. Three sessions a week for six weeks was the duration of the intervention. Standardized instruments such as the Menopause Ratings Scale (MRS) for vasomotor complaints, the severity index for insomnia (ISI), and the menu menopausal particular aspects of life and post-intervention evaluations were used to measure outcomes. The effectiveness of the measures was then compared."

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged between 45 and 60 years
* Women experiencing insomnia, vasomotor symptoms (e.g., hot flashes), and reduced quality of life
* Women who are at least 12 months amenorrheic
* Willing to participate and provide informed consent
* Physically able to perform stretching exercises

Exclusion Criteria:

* Women on hormone replacement therapy or other medications affecting sleep or menopause symptoms
* History of recent surgery or musculoskeletal injuries preventing physical activity
* Diagnosed psychiatric or neurological disorders
* Severe systemic illnesses (e.g., uncontrolled diabetes, cardiovascular diseases)
* Participation in another clinical trial or intervention in the last 3 months

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 6 Month
  insomnia. Each item is rated from 0 (no problem) to 4 (very severe problem). Total Score Range: 0-28
  0-7: No clinically significant insomnia 8-14: Subthreshold insomnia 15-21: Moderate insomnia 22-28: Severe insomnia
Menopause Rating Scale (MRS) | 6 Months
  Assesses 11 common menopausal symptoms divided into three subscales: somatic, psychological, and urogenital. Each symptom is rated from 0 (none) to 4 (very severe).
  Total Score Range: 0-44 Higher scores indicate more severe symptoms
Menopause-Specific Quality of Life Questionnaire (MENQOL) | 6 months
  A 29-item self-report scale that measures the impact of menopause on quality of life in four domains:
  Vasomotor (3 items) Psychosocial (7 items) Physical (16 items) Sexual (3 items) Each item is scored from 0 (not at all bothered) to 6 (extremely bothered). Higher scores indicate greater symptom burden and lower quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Javaid poly clinic, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No